CLINICAL TRIAL: NCT04034953
Title: Prevention of Obesity-related Cancers: Setting up of a Multi-Cancer Education and Prevention Program in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joseph JY SUNG, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: MCP Study
Record Dates: First submitted 2019-04-16; First posted 2019-07-29 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Obesity; Colorectal Cancer; Prostate Cancer; Breast Cancer
Keywords: Cancer Screening; Colorectal Cancer; Breast Cancer; Prostate Cancer; Obesity; Obesity-related Cancer; Multi-Cancer Screening
MeSH Terms: conditions — Obesity; Colorectal Neoplasms; Prostatic Neoplasms; Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colorectal Cancer Screening (Other): Potential screening participants will firstly be briefed about the CRC screening pilot program launched by the Department of Health (DH).
  This project will offer screening referrals to the government pilot program or FIT screening tests for a total of 10,000 consecutive visitors.
  Interventions: Diagnostic Test: Faecal Immunochemical Test
- Prostate Cancer Screening (Other): A blood test for Prostate Specific Antigen (PSA) will then be performed. Subsequently, for subjects with serum PSA 4-10 ng/ml, additional blood tests for Prostate Health Index (PHI) will be performed for the further assessment of risk of prostate cancer. Subjects with serum PSA > 10 ng/ml; or PHI ≥ 35 will be referred for Trans-rectal Ultrasound-guided Prostatic Biopsy (TRUS+PB). Subjects with serum PSA < 4 ng/ml or with PHI level < 35 will be invited to repeat the prostate screening tests every 2-years. We aim to screen not more than 5,000 subjects. For all patients recruited for prostate cancer screening, the study team will continue follow the subjects, by phone or mail or other means, for the long term clinical outcome for up to 10 years.
  Interventions: Diagnostic Test: Prostate-Specific Antigen Test
- Breast Cancer Screening (Other): Up to 5,000 eligible female subjects will receive a mammography on a 2-yearly basis. Individuals with abnormal findings on mammography will be referred for subsequent follow-up by the Jockey Club Breast Health Centre (BHC) run by the Hong Kong Breast Cancer Foundation (HKBCF).
  Interventions: Diagnostic Test: Mammogram

INTERVENTIONS:
Diagnostic Test: Faecal Immunochemical Test — Faecal Immunochemical Test detects if there is any hemoglobin presents in stools, so even tiny amount of blood in stool can be found.
  Other Names: FIT
  Arms: Colorectal Cancer Screening
Diagnostic Test: Prostate-Specific Antigen Test — PSA blood test is used to measure the level of PSA in blood. When the PSA level is higher than normal, it may represent prostate cancer or benign prostate hyperplasia. Patient who have high PSA level should receive additional tests.
  Other Names: PSA
  Arms: Prostate Cancer Screening
Diagnostic Test: Mammogram — Each sides of breast will be taken imaging in 2 different views.The breast will be pressed between 2 plastic plates to flatten and spread the breast tissue for clear imaging.
  Other Names: MMG
  Arms: Breast Cancer Screening

SUMMARY:
Obesity could increase the risk of many chronic diseases, including hypertension, cardiovascular diseases, high lipid level, diabetes, stroke, endometrial cancer and certain types of cancer which could benefit by secondary prevention through screening programs. The World Cancer Research Fund of the American Institute for Cancer Research has reviewed all the studies about the link between obesity and cancer. Studies shown that obesity is an independent risk factor for colorectal, breast and prostate cancer. These three cancers (will be named as "obesity-related cancers" thereafter) demonstrate a rapidly increasing trend of incidence in Asia in the past decade.

Among Chinese adults of Hong Kong in 2014, 39% were overweight or obese (compared with 20.9% reported in European adults in the same year) and up to 69.7% reported that they did not perform any measures to achieve optimal weight control. Men (49.6%) had a higher proportion of overweight or obesity than females (29.5%). Adults who are aged 45-54 had the highest rate (50.5%) of overweight or obesity than other age groups. In addition, there were 62.5% whose physical activity level did not meet the recommendations from the World Health Organization (WHO). Only 18.7% consumed at least 5 portions of fruit and vegetables per day; yet about 30% were alcoholic drinkers; and more than 10% were daily or occasional smoker. These figures imply that the incidence of obesity and obesity-related cancers will further escalate - and urgent actions at the community level are needed to combat the rising incidence and mortality of these conditions.

According to Hong Kong Cancer Registry, the discrepancy between the number of new cases (incidence) and number of deaths (mortality) is much higher for colorectal, breast and prostate cancer as compared to other cancers. It is well recognized that screening could effectively reduce mortality for these three obesity-related cancers when they are detected at an earlier stage.

The concept of a one-stop approach to screen for multiple cancers was found to be feasible, with an ability to detect a wide range of neoplastic lesions at an early stage. In the recent decade, there are also emerging centres that have been established as multi-cancer screening clinics worldwide. Nevertheless, there is a scarcity of studies that have highlighted the outcomes of these multi-cancer screening programs.

DETAILED DESCRIPTION:
Obesity could increase the risk of many chronic diseases, including hypertension, cardiovascular diseases, high lipid level, diabetes, stroke, endometrial cancer and certain types of cancer which could benefit by secondary prevention through screening programs. In particular, colorectal, breast and prostate cancer (these three cancers will be named as "obesity-related cancers" thereafter) demonstrate a rapidly increasing trend of incidence in Asia in the past decade. The World Cancer Research Fund of the American Institute for Cancer Research has reviewed all the studies about the link between obesity and cancer . For colorectal cancer (CRC), there is compelling evidence suggesting that obesity is associated with 30-66% higher risk of developing CRC. Weight gain during adulthood was also shown to increase risk of CRC. As for breast cancer, post-menopausal women with the smallest waist (compared with the largest) had 39% lower risk of getting breast cancer . A 5-unit increase in BMI is associated with 12% increased risk of breast cancer, and this figure escalates to 20-40% for postmenopausal women. For prostate cancer, greater body fatness has been suggested as a reason of advanced prostate cancer. Obesity was positively related to advanced stage prostate cancer. The relative risk is 1.09 for every 5 kg/m2 higher BMI.

Among Chinese adults of Hong Kong in 2014, 39% were overweight or obese (compared with 20.9% reported in European adults in the same year) and up to 69.7% reported that they did not perform any measures to achieve optimal weight control. Men (49.6%) had a higher proportion of overweight or obesity than females (29.5%). Adults who are aged 45-54 had the highest rate (50.5%) of overweight or obesity than other age groups. In addition, there were 62.5% whose physical activity level did not meet the recommendations from the World Health Organization (WHO). Only 18.7% consumed at least 5 portions of fruit and vegetables per day; yet about 30% were alcoholic drinkers; and more than 10% were daily or occasional smoker. These figures imply that the incidence of obesity and obesity-related cancers will further escalate - and urgent actions at the community level are needed to combat the rising incidence and mortality of these conditions.

As shown in Figure 2, the discrepancy between the number of new cases (incidence) and number of deaths (mortality) is much higher for colorectal, breast and prostate cancer as compared to other cancers. It is well recognized that screening could effectively reduce mortality for these three obesity-related cancers when they are detected at an earlier stage.

Primary prevention is one of the crucial strategies found to be effective in cancer prevention. Health education on modification of lifestyle factors is especially useful to change behavior and reduce the impact of the threats posed by obesity and its related cancers. The application of behavioral medicine, defined as "the interdisciplinary field concerned with the development and integration of sociocultural, psychosocial, behavioral, and biomedical knowledge relevant to health and illness and the application of this knowledge to disease prevention, health promotion, etiology, diagnosis, treatment, and rehabilitation'', has been considered to be the most effective and practical means to prevent cancers. A comprehensive strategy for reducing cancers also includes secondary prevention that aims at early detection of diseases. Early detection for some "screen-relevant" cancers is particularly effective to reduce cancer-related mortality.

The concept of a one-stop approach to screen for multiple cancers is relatively novel from existing literature - and one of such initiatives is the "Integrated Cancer Prevention Centre" (ICPC) established in Tel Aviv Sourasky Medical Center at Israel in 2006. Analysis of the first 1,000 subjects visiting the centre showed that the compliance at the centre was higher than those seen in the Ministry of Health for the general population (78% vs. 60% for mammography; 39% vs. 16% for colonoscopy). The provision of such a unique facility designed for one-stop screening for multiple cancers was found to be feasible, with an ability to detect a wide range of neoplastic lesions at an early stage. In the recent decade, there are also emerging centres that have been established as multi-cancer screening clinics worldwide. Nevertheless, there is a scarcity of studies that have highlighted the outcomes of these multi-cancer screening programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years depending on risk factor(s);
* Measured BMI ≥ 25 kg/m2; or waist circumference >80cm [women] or >90 cm [men]; and
* Absence of existing or previous symptoms suggestive of CRC and breast cancer

Exclusion Criteria:

* Having received updated CRC screening tests (FIT in the past 2 year; flexible sigmoidoscopy in the past 5 years; colonoscopy in the past 10 years);
* Having received updated prostate or breast screening test in the past 2 years;
* Having personal of CRC, prostate or breast cancers;
* Having personal history of colonic adenoma, diverticular disease or inflammatory bowel disease;
* Having medical conditions which were contraindications for colonoscopy, like cardiopulmonary insufficiency and the use of double antiplatelets, etc.; and
* Having medical conditions and disabling conditions with limited life expectancy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Colorectal cancer detection rate | 5 Years
  Evaluate the effectiveness of CRC screening in a one-stop community based obesity-related cancers screening program
Prostate cancer detection rate | 5 Years
  Evaluate the effectiveness of prostate cancer screening in a one-stop community based obesity-related cancers screening program
Breast cancer detection rate | 5 Years
  Evaluate the effectiveness of breast cancer screening in a one-stop community based obesity-related cancers screening program

CONTACTS AND LOCATIONS:
Overall Officials: Joseph JY Sung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Lek Yuen Health Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Access to the data or study record will be available to authorized research staff (eg, Principle Investigator, Co-Investigators, research assistant, etc) only, during and after the study.

REFERENCES:
- [Derived] Zhu Z, Lam TYT, Tang RSY, Wong SH, Lui RNS, Ng SSM, Wong SYS, Sung JJY. Triglyceride-glucose index (TyG index) is associated with a higher risk of colorectal adenoma and multiple adenomas in asymptomatic subjects. PLoS One. 2024 Nov 7;19(11):e0310526. doi: 10.1371/journal.pone.0310526. eCollection 2024. PMID 39509387
- [Derived] Sung JJY, Luk AKC, Ng SSM, Ng ACF, Chiu PKF, Chan EYY, Cheung PSY, Chu WCW, Wong SH, Lam TYT, Wong SYS. Effectiveness of One-Stop Screening for Colorectal, Breast, and Prostate Cancers: A Population-Based Feasibility Study. Front Oncol. 2021 Feb 25;11:631666. doi: 10.3389/fonc.2021.631666. eCollection 2021. PMID 33718212